CLINICAL TRIAL: NCT02347059
Title: A Randomized, Single-blind Trial on the Efficacy and Safety of L-dopa Monotherapy Versus Dopamine Agonists Monotherapy After Subthalamic Nucleus Deep Brain Stimulation in Parkinson's Disease
Brief Title: L-dopa Versus Dopamine Agonists After Subthalamic Nucleus Deep Brain Stimulation in Parkinson's Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Toronto (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Principal Investigator, Alfonso Fasano, Associate Professor, Movement Disorders centre, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-8303
Record Dates: First submitted 2015-01-20; First posted 2015-01-27 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Levodopa; Dopamine Agonists; Pramipexole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- L-dopa (Experimental): L-dopa will be administered as monotherapy. The dosage and the frequency of intakes are not pre-specified and will be individualized.
  Interventions: Drug: L-dopa
- Dopamine agonist (Active Comparator): Dopamine agonists (either pramipexole or ropirinole) will be administered as monotherapy. The dosage and the frequency of intakes are not pre-specified and will be individualized.
  Interventions: Drug: Dopamine Agonists (pramipexole, ropirinole)

INTERVENTIONS:
Drug: L-dopa — Antiparkinsonian medication
  Other Names: Levodopa
  Arms: L-dopa
Drug: Dopamine Agonists (pramipexole, ropirinole) — Antiparkinsonian medication
  Other Names: Pramipexole; Ropirinole
  Arms: Dopamine agonist

SUMMARY:
Deep Brain Stimulation (DBS) of the Subthalamic nucleus (STN) is an established treatment for patients with advanced Parkinson's disease (PD). STN DBS improves dopaminergic drug-responsive motor symptoms, thus allowing a reduction of post-operative drug dose. However, a considerable variation in the extent of dopaminergic drug reduction has been reported, with values ranging from 20% to 100%. Both L-dopa and DAs can be used, however, there are no formal studies examining which type of antiparkinsonian medication may be more effective and/or better tolerated following STN DBS.

Aim of our study is to compare the efficacy and the tolerability of L-dopa monotherapy versus DAs monotherapy after STN DBS over a 3-month follow up period.

This study is a prospective, single blind parallel trial comparing L-dopa monotherapy and DAs monotherapy after STN DBS. Patients will be enrolled in pairs, with one patient randomly assigned to L-dopa monotherapy and the other to DA monotherapy after STN DBS (20 patients for each study arm). Treatment assignment will be unmasked for the patient but will be blinded for the neurologist programming DBS and evaluating the patient. Another neurologist will be in charge of medication adjustments. Primary outcome is the change in severity of non-motor symptoms as assessed by the Non-motor Symptoms Scale (NMSS) at 3-month follow up visit after surgery.

In spite of an improvement of the motor condition many patients develop apathy and depression following surgery ("Neurosurgery in Parkinson's disease: the doctor is happy, the patient less so"). This study will shed light on the best way to manage patients after STN procedure, thus contributing to a further improvement of the surgical outcome in a population of young and motivated patients (those commonly receiving STN DBS), eventually bringing them closer to a normal personal and social life.

Results of our study may provide new insights in the management of advanced PD after STN DBS, further leading to development of future larger trials.

DETAILED DESCRIPTION:
Background Information Deep Brain Stimulation (DBS) of the Subthalamic nucleus (STN) is an established treatment for patients with advanced Parkinson's disease (PD). STN DBS improves dopaminergic drug-sensitive motor symptoms, thus allowing a reduction in post-operative drug dose. The reduction of antiparkinsonian therapy in turn alleviates L-dopa-induced motor fluctuations and dyskinesias. However, a considerable variation in the extent of dopaminergic drug reduction has been reported, with values ranging from 20% to 100%. To date the management of antiparkinsonian medication after STN DBS mainly rely on neurologist's personal experience or patient's preference, as no evidence-based guidelines have been provided so far, with the exception of some pragmatic recommendation on postoperative issues promoted by the Movement Disorders Society in 2006.

Rationale for the study, potential risks and benefit In the immediate postoperative period following STN DBS, simplification of the medication regimen is advised, given the complexity of the interactions between stimulation and medication. Both L-dopa and DAs can be used, however, there are no formal studies examining which type of antiparkinsonian medication may be more effective and/or better tolerated following STN DBS. In spite of the need of simplification of the medication regimen after STN DBS in PD, to date there are no clinical trials specifically designed to compare the efficacy (in terms of motor and non-motor outcomes) and safety of L-dopa monotherapy versus DAs monotherapy following STN DBS.

Description of the population to be studied Patients with Parkinson's disease in advanced stage who undergo STN DBS. After one months since surgery, during the first programming visit, patients will be randomized in two groups receiving either L-dopa monotherapy or DAs monotherapy (either with pramipexole or ropirinole) for 2 months.

Study objectives and hypothesis Aim of our study is to compare the efficacy and the safety of L-dopa monotherapy versus DAs monotherapy after STN DBS over a 3-month follow up period. The hypothesis is that DAs may be more efficacious than L-dopa in treating non-motor symptoms after surgery, thus further improving quality of life following surgery. On the other hand, in comparison with L-dopa, DAs might be associated with more side effects (in particular impulse control disorders) and less effective motor control.

Study design This study is a prospective, single blind trial with a randomized-pairs design comparing L-dopa monotherapy and DAs monotherapy after STN DBS. The trial will be a single-center pilot study, conducted at Toronto Western Hospital, Toronto, Canada. The protocol meets the Ethical Conduct for Research Involving Humans. All patients will provide written informed consent. A total of 40 patients is estimated to be enrolled (20 patients for each treatment group). Duration of the study is 15 months. Enrollment will last for 12 months. The center will enroll patients in pairs, with one patient randomly assigned to L-dopa monotherapy and the other to DAs monotherapy after STN DBS. Randomization will be performed generating a random sequence of number through block randomization. Treatment assignment will be unmasked for the patient but will be blinded for the neurologist programming DBS and evaluating the patient. Another neurologist will be in charge of medication adjustments. Randomization, monitoring, and data management and analysis will be performed at the Toronto Western Hospital.

Selection of subjects Subjects will be screened while they perform the standard pre-operative assessments (including a videotaped L-dopa challenge, a psychiatric evaluation, neuropsychological assessment and the visit with the neurosurgeon). If they are treated with both L-dopa and DAs (either pramipexole or ropirinole) prior to surgery they will be asked to participate in the study. If they accept, they will undergo the first visit (about one month before surgery). During the first visit they will be administered scales and questionnaires evaluating both your motor and non-motor symptoms (i.e. apathy, mood, sleep) related to Parkinson's disease. This evaluation will last about 1 hour. Then, enrolled subjects will undergo surgery according to the standard of practice currently adopted at Toronto Western Hospital. For the first month after surgery their medication will be unchanged. After one month since surgery they will have their first programming visit. During this visit, enrolled subjects will be randomized either to join the L-dopa group or the DAs group (receiving either pramipexole or ropirinole).

Study Interventions Bilateral simultaneous STN implants will be performed in all patients using the standard stereotactic technique adopted at Toronto Western Hospital. According to the standard of practice currently adopted at Toronto Western Hospital, DBS patients will undergo a pre-surgical evaluation (including a videotaped L-dopa challenge to verify the response of motor symptoms to L-dopa, a neuropsychological evaluation, a psychiatric assessment and a visit with the neurosurgeon). Then, they will be seen one month after surgery for the first programming visit (when the "microlesional" effect is supposed to be gone) and then once a week for the subsequent 8 weeks (in order to slowly adjusts DBS parameters). The optimal stimulation settings will be progressively adjusted according to the patient's response. The standard pulse setting will be 60 μsec in duration at 130 Hz, with voltage adjusted to the individual patient. As regards antiparkinsonian treatment, patients will be randomly assigned to L-dopa monotherapy or DAs monotherapy during the first programming visit. During the 8-weeks adjustment period, L-dopa or DAs (depending on the study arm) will be slowly tapered off and dose of the drug left in monotherapy will be adjusted according to the patient's clinical condition. According to the standard of practice, the drugs dosage will be adjusted according to the patient's needs and will be maintained to the minimum sufficient level to achieve optimal motor control in absence of side effects throughout the duration of the study. In keeping with the standard of care at Toronto Western, patients will then be seen after 3 months since surgery for the completion of the study visit. However, unscheduled visits will be possible in case of unexpected clinical conditions (i.e. occurrence of side effects or worsening of motor conditions).

L-dopa and DAs (both pramipexole and ropirinole) are very well known drugs, commercially available and approved for treatment as monotherapy and as adjunct therapy for Parkinson's disease in Canada by the Terapeutic Products Directorate of Health Canada. All potential side effects will be actively monitored through the study.

The total length of the study is 15 months. First, the patients will be screened as to your suitability for this study. This will happen while the patients are performing the standard pre-operative assessments (including a videotaped L-dopa challenge, a psychiatric evaluation, neuropsychological assessment and the visit with the neurosurgeon). If the surgical candidates are treated with both L-dopa and DAs (either pramipexole or ropirinole) prior to surgery they will be asked to participate in the study. If they accept, they will undergo the first visit (about one month before surgery). During the first visit they will be administered scales and questionnaires evaluating both your motor and non-motor symptoms (i.e. apathy, mood, sleep) related to Parkinson's disease. This evaluation will last about 1 hour. Then, the patients will undergo surgery according to the standard of practice currently adopted at Toronto Western Hospital. For the first month after surgery their medication will be unchanged. After one month since surgery the patients will have your first programming visit. During this visit, the enrolled patients will be randomized either to join the L-dopa group or the DAs group (receiving either pramipexole or ropirinole). If they will be assigned to the L-dopa group you will gradually discontinue DAs, while if they will be randomized to join the DAs group you will gradually discontinue L-dopa. Then, every patient will be seen once a week for the subsequent 8 weeks to optimize both the stimulations settings and the medical treatment. After 3 month since surgery the enrolled patients will have the last visit of the study and will receive the same scales and questionnaires evaluating both your motor and non-motor symptoms (i.e. apathy, mood, sleep) related to Parkinson's disease. This evaluation will again last about 1 hour.

Throughout the study the patients will perform approximately 9-11 visits, according to the standard of practice currently adopted at Toronto Western Hospital. All evaluations will be conducted in the outpatient clinic. The assessments relative to this study will be administered to enrolled subjects twice (once during the pre-surgical assessments and again during the 3-month follow up visit). Safety and tolerability will be assessed by recording the frequency and the severity of reported adverse events during each visit.

Statistical analysis The impact of STN DBS on non-motor symptoms of PD has not been extensively studied and only limited data are available. Based on these data, we anticipate that in order to detect a between-group change of the Non-motor Symptoms Scale (NMSS) of at least 23.3 points the sample size should be of at least 20 patients per each study arm, assuming a power of 0.80 and an alpha value of 0.05. Such a difference is not as large as it seems as the NMSS total score ranges from 0 to 360. Furthermore, this estimation was computed on a pilot study with a small sample size. Beyond that, the NMSS also includes a subscore for each of the 9 domains. Those will be analyzed as well. Presurgical differences between treatment groups will be evaluated with parametric or non-parametric tests, as appropriate. Mean changes in the continuous variables between baseline and 3-month follow up after STN DBS will be compared within and between treatment groups using repeated measures analysis of variance with "treatment group" and "time" as independent categorical factors. The interactions between dependent variables and any other variable of interest (e.g. age, MDS-UPDRS-III, stimulation parameters) will be entered into the model. Given the nature of our study, the standard non corrected significance α level of p<0.05 will be used.

Direct access to Source/Data Documents Reasonable access to study data will be provided to the funder (The Michael J. Fox Foundation for Parkinson's research, MJFF) in a format prescribed by it (defined as one or all of the following: the final clinical study report, final clinical datasets and listing that have been de-identified according to the HIPAA and its implementing regulations). MJFF, its grant assessors, and MJFF consultants will use such information only internally to make future funding decisions. MJFF shall have the right to audit and review detailed data related to the project.

Quality control and quality assurance procedures All clinical trial information will be recorded, handled, and stored in a way that allows its accurate reporting, interpretation, and verification. Systems with procedures that assure the quality of every aspect of the trial will be implemented (i.e. check list). Quality control will be applied to each stage of data handling to ensure that all data are reliable and have been processed correctly.

ELIGIBILITY:
Inclusion Criteria:

1. patients with a clinical diagnosis of idiopathic PD according to the British Parkinson's Disease Society Brain Bank criteria
2. medical treatment with both L-dopa and DAs (either pramipexole or ropirinole) prior to surgery
3. candidacy for STN DBS according to the treating physician and fulfillment of the inclusion and exclusion criteria proposed by the core assessment program for surgical interventional therapies in Parkinson's disease panel
4. Informed consent to participate in the study

Exclusion Criteria:

* History of active ICDs or depression (according to internal and international guidelines these patients are not deemed as surgical candidate)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Severity at 3-month follow up visit after surgery of non-motor symptoms as assessed by the Non-motor Symptoms Scale (NMSS) | 3 months

SECONDARY OUTCOMES:
activities of daily living as assessed by the MDS Unified Parkinson's Disease Rating Scale, Activities of daily living section (MDS-UPDRS-II) | 3 months
• the severity of motor symptoms, as assessed by the MDS Unified Parkinson's Disease Rating Scale, motor section (MDS-UPDRS-III) | 3 months
• motor fluctuations and dyskinesias as assessed by the MDS Unified Parkinson's Disease Rating Scale, part IV (MDS- UPDRS-IV) | 3 months
• the quality of life, as assessed by the Parkinson's Disease Questionnaire (PDQ-39) summary index | 3 months
• prevalence and severity of depression and apathy as assessed by the Hospital Anxiety Depression Scale (HADS) and the Apathy Evaluation Scale (AES, both self- and informant-rating scales) | 3 months
• severity and occurrence of ICDs, as rated with the Questionnaire for Impulsive-Compulsive Disorders in Parkinson's Disease (QUIP scale) | 3 months
• severity and occurrence of sleep disorders, as rated with the Parkinson's disease Sleep Scale (PDSS) | 3 months
Safety and tolerability will be assessed by recording the frequency and the severity of reported adverse events during each visit. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Alfonso Fasano, MD, PhD, Principal Investigator — Movement Disorders Centre Toronto Western Hospital
Locations (1):
- Movement disorders Centre, Toronto Western Hospital, Toronto, Ontario, Canada